CLINICAL TRIAL: NCT05829226
Title: A Phase 1 Open-label, Multi-center Study of the Safety, Pharmacokinetics (PK), and Anti-tumor Activity of LYT- 200 in Patients With Relapsed/Refractory Acute Myeloid Leukemia (AML), or With Relapsed/Refractory, High-risk Myelodysplastic Syndrome (MDS)
Brief Title: A Phase 1 Study With LYT-200 in Patients With Relapsed/Refractory Acute Myeloid Leukemia (AML), or With Relapsed/Refractory, High-risk Myelodysplastic Syndrome (MDS)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: PureTech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LYT-200-2022-02
Record Dates: First submitted 2023-03-30; First posted 2023-04-25 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: AML, Adult Recurrent; MDS
Keywords: AML Recurrent; AML Relapsed; AML Refractory; Hematological Cancer; Gal-9; Immuno-oncology; MDS; MDS High Risk
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — venetoclax; Azacitidine; Decitabine

STUDY DESIGN:
Intervention Model Description: A Phase 1 open-label, multi-center study. The 4+2 algorithm-based dose-escalation design in single agent LYT-200 and in combination with venetoclax and/or HMAs will be used to help identify the recommended Phase 2 dose (RP2D). Up to 6 patients per single treatment Cohorts 1-5 will receive infusions of LYT-200 every week (QW). Up to 6 patients per combination Cohorts 1-4 will receive infusions of LYT-200 QW and oral venetoclax every day and/or HMAs for 7 days (azacitidine) or 5 days (decitabine) per cycle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single agent dose escalation (Experimental): LYT-200 in relapsed/refractory AML or relapsed/refractory high-risk MDS, administered via IV infusion over 60 minutes every week.
  Interventions: Drug: LYT-200
- Combination agent dose escalation (Experimental): LYT-200 in relapsed/refractory AML or relapsed/refractory high-risk MDS, administered via IV infusion over 60 minutes every week, in combination with oral venetoclax Day 1, 100 mg, Day 2, 200mg, Day 3-28, 400 mg and/or azacitidine, 75 mg/m2 subcutaneously given for 7 days per cycle or decitabine 20 mg/m2 IV for 5 days per cycle.
  Interventions: Drug: LYT-200; Drug: Venetoclax; Drug: Azacitidine; Drug: Decitabine

INTERVENTIONS:
Drug: LYT-200 — monoclonal antibody (mAb), targeting galectin-9 protein
Drug: Venetoclax — Bcl-2 inhibitor
  Arms: Combination agent dose escalation
Drug: Azacitidine — Hypomethylating agent
  Arms: Combination agent dose escalation
Drug: Decitabine — Hypomethylating agent
  Arms: Combination agent dose escalation

SUMMARY:
A Phase 1 Open-label, Multi-center Study of the Safety, Pharmacokinetics (PK), and Anti-tumor Activity of LYT- 200 in Patients with Relapsed/Refractory Acute Myeloid Leukemia (AML), or with Relapsed/refractory, High-risk Myelodysplastic Syndrome (MDS)

DETAILED DESCRIPTION:
This is an open-label, non-randomized, multi-center, Phase 1, dose escalation study in patients with AML relapsed/refractory to at least one line of prior therapy, with or without an allogeneic stem cell transplant, or in patients with a documented diagnosis of relapsed/refractory, high-risk myelodysplastic syndrome (MDS) post at least one line of treatment and for whom no standard therapy that may provide clinical benefit is available. The 4+2 algorithm-based dose-escalation design will be used to help identify the recommended Phase 2 dose (RP2D). Single agent LYT-200 and in combination with venetoclax and/or hypomethylating agents (HMA) safety and tolerability evaluation is the primary study endpoint, Pharmacokinetics (PK), and Anti-tumor Activity of LYT- 200 single agent and in combination with venetoclax and/or HMAs are key secondary study endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age at the time of obtaining informed consent.
* Patients with morphologically documented primary or secondary AML by the World Health Organization(WHO) criteria, whose disease is relapsed/refractory to at least one line of prior therapy, with or without an allogeneic stem cell transplant and for whom no standard therapy that may provide clinical benefit is available or for patients who decline available standard of care.
* Patients with a documented diagnosis of high-risk myelodysplastic syndrome (MDS), whose disease is relapsed/refractory, post at least one line of treatment based on the revised International Prognostic Scoring System (IPSS-R) and for whom no standard therapy that may provide clinical benefit is available
* Patients are able and willing to comply with study procedures as per protocol, including bone marrowbiopsies.
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Patient must meet the following criteria as indicated on the clinical laboratory tests:

oWhite blood cell (WBC) count at the time of the first dose of < 25,000/uL. oAspartate aminotransferase or alanine aminotransferase ≤ 3 × upper limit of normal (ULN; ≤ 5.0× ULN if considered to be due to leukemic involvement). oTotal bilirubin ≤ 2 × ULN (≤ 3 × ULN if considered to be due to leukemic involvement orGilbert's syndrome). oCreatinine clearance of ≥ 60 mL/min.

Exclusion Criteria:

* Patient diagnosed with acute promyelocytic leukemia (APL).
* Patient has active malignant tumors other than AML/MDS
* Patient has had HSCT and meets any of the following: has undergone HSCT within the 6- month period prior to the first study dose; has ≥ Grade 2 persistent non-hematological toxicity related to the transplant donor lymphocytes infusion.
* Patient has active graft versus host disease (GVHD) and patients receiving immunosuppressive treatment for GVHD.
* Patient with symptomatic central nervous system (CNS) involvement of leukemia or other CNS diseases related to underlying and secondary effects of malignancy
* Patient has had major surgery within 4 weeks prior to the first study dose.
* Patient has congestive heart failure New York Heart Association (NYHA) class 3 or 4, or patient with a history of congestive heart failure NYHA class 3 or 4 in the past, unless a screening echocardiogram or multigated acquisition (MUGA) scan performed within 3 months prior to study entry results in a left ventricular ejection fraction (LVEF) that is ≥ 45%.
* Patient has any condition which, in the Investigator's opinion, makes the patient unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and RP2D determination] | approximately 1 year
  Evaluation of safety parameters including treatment emergent adverse events as detected by hematology, chemistry, coagulation safety labs, physical exams, vital signs, ECG, ECHO/MUGA, ECOG status
Incidence of Dose Limiting Toxicities [Tolerability and RP2D determination] | approximately 1 year
  Evaluation of tolerability parameters including dose limiting toxicities as detected by hematology, chemistry, coagulation safety labs, physical exams, vital signs, ECG, ECHO/MUGA, ECOG status

SECONDARY OUTCOMES:
Rate of disease responses, time-to-event endpoints, hematological improvements | approximately 1 year
  Evaluate preliminary efficacy of LYT- 200 as a single agent in AML and MDS
Pharmacokinetic (PK) profile of LYT-200_Area Under the Curve (AUC) | approximately 1 year
  Characterize the PK profile of LYT-200
Pharmacokinetic (PK) profile of LYT-200_Concentration Max (CMax) | approximately 1 year
  Characterize the PK profile of LYT-200
Pharmacokinetic (PK) profile of LYT-200_Time to Reach CMax (TMax) | approximately 1 year
  Characterize the PK profile of LYT-200

OTHER OUTCOMES:
Anti-Drug Antibody formation | approximately 1 year
  Assess the immunogenicity of LYT-200

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Filipovic, MD, PhD., Study Director — PureTech Health
Locations (9):
- United States (9):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Irvine Medical Center, Orange, California
  - Baptist Health South Florida-Miami Cancer Institute, Miami, Florida
  - Norton Healthcare-Norton Cancer Institute, Louisville, Kentucky
  - Mass. General Hospital-Harvard, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rhode Island Hospital, Providence, Rhode Island
  - Virginia Commonwealth University Medical Center, Richmond, Virginia